CLINICAL TRIAL: NCT04439864
Title: Perspectives Post Percutaneous Coronary Intervention Randomized Study
Brief Title: Perspectives Patient Education Randomized Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Cook County Health (Other Government); National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Andrew D Boyd, Association Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 2013-0802; P30AG022849 (NIH); UL1TR000050 (NIH); P30NR010680 (NIH)
Record Dates: First submitted 2020-06-11; First posted 2020-06-19 (Actual); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: Medication Adherence
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MyIDEA (Experimental): Research Participants interacted with MyIDEA program both in the hospital and in the follow up cardiology appointment.
  Interventions: Device: MyIDEA
- Treatment as normal (No Intervention): The research participants were given the chance to play games on the tablet and received normal clinical education.

INTERVENTIONS:
Device: MyIDEA — An educational tablet app that is customized to the patient based on the data in the Electronic Health Record.
  Arms: MyIDEA

SUMMARY:
This is a randomized clinical trial evaluating the educational program called My Interventional Drug Eluting Stent Educational App (MyIDEA) that is a pilot at two sites.

ELIGIBILITY:
Inclusion Criteria:

1. received a drug eluting stent during a Percutaneous Coronary Intervention (PCI) during a hospitalization for the PCI procedure,
2. were greater than 50 years old (funding agency requirement),
3. spoke and understood English.

Exclusion Criteria:

1. inability to give informed consent
2. allergy to aspirin

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-05-01 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
Feasibility of study design engaging elderly patients in novel tablet based education. | 3 months
  Would research participants enroll and follow up in a study of tablet based education. Do patients think they know everything? Would patients enrolled in the control arm still follow up in the study?

SECONDARY OUTCOMES:
Medication adherence | 3 months
  A measure of Pharmacy days covered for DAPT medication. The patients after recieving a Drug Eluting Stent need to adhere to Dual Antiplatlet Therapy (DAPT) to prevent restenosis of the stent. PDC is a calculation of the DAPT which is Aspirin and an ADP receptor antagonist. As aspirin is over the counter, the pharmacy does not have a record of purchase so the PDC was calculated for the ADP receptor antagonis.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew D Boyd, MD, Principal Investigator — University of Illinois at Chicago

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shah V, Dileep A, Dickens C, Groo V, Welland B, Field J, Baumann M, Flores JD, Shroff A, Zhao Z, Yao Y, Wilkie DJ, Boyd AD. Patient-Centered Tablet Application for Improving Medication Adherence after a Drug-Eluting Stent. Front Public Health. 2016 Dec 12;4:272. doi: 10.3389/fpubh.2016.00272. eCollection 2016. PMID 28018897
- [Result] Boyd AD, Moores K, Shah V, Sadhu E, Shroff A, Groo V, Dickens C, Field J, Baumann M, Welland B, Gutowski G, Flores JD Jr, Zhao Z, Bahroos N, Hynes DM, Wilkie DJ. My Interventional Drug-Eluting Stent Educational App (MyIDEA): Patient-Centered Design Methodology. JMIR Mhealth Uhealth. 2015 Jul 2;3(3):e74. doi: 10.2196/mhealth.4021. PMID 26139587
- [Derived] Boyd AD, Ndukwe CI, Dileep A, Everin OF, Yao Y, Welland B, Field J, Baumann M, Flores JD Jr, Shroff A, Groo V, Dickens C, Doukky R, Francis R, Peacock G, Wilkie DJ. Elderly Medication Adherence Intervention Using the My Interventional Drug-Eluting Stent Educational App: Multisite Randomized Feasibility Trial. JMIR Mhealth Uhealth. 2020 Jun 24;8(6):e15900. doi: 10.2196/15900. PMID 32579120